CLINICAL TRIAL: NCT01733160
Title: SPRINT-AF: Stroke Prevention and Rhythm Interventions in Atrial Fibrillation
Brief Title: Stroke Prevention and Rhythm Interventions in Atrial Fibrillation
Acronym: SPRINT-AF
Status: Completed | Type: Observational
Sponsor: Canadian Collaborative Research Network (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: SPRINT-AF 18-10-2012
Record Dates: First submitted 2012-11-02; First posted 2012-11-26 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Diseases
Keywords: Atrial Fibrillation; Stroke; Anticoagulants
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational registry will characterize contemporary stroke prevention in Canadian adults with atrial fibrillation, and provide clarity in understanding physician preferences for the various oral anticoagulants available in the Canadian marketplace. This study will determine the patient profiles of those selected for the various therapies available in Canada and provide an understanding of the factors involved in drug selection and management.

DETAILED DESCRIPTION:
Atrial fibrillation affects approximately 1% of the general population, and the prevalence of AF increases with increasing age, such that 10-15% of individuals aged 80 years or greater suffer from AF. Various projections estimate at least a doubling of the prevalence of AF over the next 30-40 years. Stroke is a serious, often disabling complication of AF. The Framingham Heart Study demonstrates a roughly five-fold increase in the risk of stroke in patients with AF. The proportion of strokes attributable to AF also increases with age, such that one quarter to one third of all strokes in octogenarians are related to atrial fibrillation.

AF-related strokes tend to be more severe than ischemic strokes of other etiologies, resulting in a higher rate of stroke-related disability. Vitamin K antagonists have been shown to be highly effective in reducing the risk of stroke in patients with AF. A recent meta-analysis of 6 trials of VKA versus placebo, in over 2900 patients with AF, demonstrated a roughly 65% reduction in thromboembolic stroke. Thus, vitamin K antagonists (VKA) have been universally recommended for most AF patients felt to be at moderate to high risk for stroke. The CHADS2 risk score fairly accurately distinguishes patients at low, moderate and high risk for stroke using clinical variables in a bedside risk score. In recent years, VKA have been recommended for AF patients with a CHADS2 risk score of at least 2 or greater, with the optional use of either ASA or VKA for those with a score of 1. Most recently, the Canadian Cardiovascular Society's 2010 AF Guidelines now recommend anticoagulation for patients with a CHADS2 risk score of 1 or greater, in the absence of increased bleeding risk. The 2012 update to the Canadian Cardiovascular Society Guidelines additionally recommends the use of the CHA2DS2-Vasc score in patients with a CHADS2 risk score of 0, and subsequent use of OAC even in a proportion of these patients.

The benefits of VKA are largely dependent upon achieving adequate anticoagulation, ideally an INR of between 2 and 3, for the majority of treatment time. However, achieving and maintaining therapeutic anticoagulation in clinical practice can be quite challenging. Warfarin and other VKA have a variety of limitations in clinical practice. The individual patient's response to warfarin is often unpredictable, with a narrow therapeutic window. The drug has a slow onset and offset of action, with the need for regular INR monitoring and frequent dose adjustments. There are often numerous food and drug interactions with warfarin. Patients may be non-compliant with routine INR monitoring. Physicians may be wary of the risk of bleeding complications, particularly the risk of intracranial haemorrhage, which rises substantially once INR approaches 4 or beyond. Such fear of bleeding may lead physicians to underprescribe warfarin to patients at increased stroke risk. Adverse events with warfarin are common, leading to a high rate of discontinuation. As a result of these limitations, it is estimated that only half of eligible AF patients worldwide receive any VKA at all. In those patients receiving VKA, only 40-60% actually achieve therapeutic anticoagulation. The adequacy of anticoagulation with VKA is often termed "Time in Therapeutic Range (TTR)", which estimates the overall period of time that an individual patient or group of patients spend with an INR between 2 and 3. Numerous practice audits and observational registries suggest that the average TTR globally is roughly 45-55%, whereas it is estimated that a TTR of 65% is required to optimally reduce the risk of AF-related stroke.

In addition, a variety of other issues must be considered in the management of patients with AF, such as rate vs. rhythm control, drug selection, device therapy, and management of associated co-morbidities, in particular, hypertension.

Recently, two new classes of oral anticoagulants have entered the Canadian marketplace. These include dabigatran, a direct thrombin inhibitor, and rivaroxaban, a factor Xa inhibitor. Both drugs offer distinct advantages over warfarin, provide predictable anticoagulation without the need for monitoring, and have different safety and tolerability profiles. It is unknown how Canadian physicians currently assess and manage stroke risk in patients with AF, and it is also unknown how physicians will adopt new oral anticoagulants into their practices. Recent guidelines also highlight the need for physicians to assess bleeding risk in AF patients, something that most physicians do not perform in a systematic manner. Thus, in this new era of stroke prevention strategies and guidelines, a prospective AF registry is clearly warranted to better understand physician approaches to the use of OAC in clinical practice, and to characterize patient variables determining the use of specific agents.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation (ECG, rhythm strip, device interrogation, discussion of an AF diagnosis in the participant's clinical report) within the past 10 years; paroxysmal, persistent or permanent
* Age > 18 years
* Most recent visit for a patient having had a clinical visit with Investigator occurring within the past one year

Exclusion Criteria:

* Valvular AF (hemodynamically significant valvular heart disease including rheumatic mitral valve disease or at least moderate aortic valve stenosis)
* Life expectancy < 12 months
* Active malignancy (treated or untreated)
* Indication for systemic anticoagulation independent of atrial fibrillation (venous thromboembolism, mechanical heart valve)
* Prior participation in any OAC randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care and specialist clinics
Sampling Method: Probability Sample
Enrollment: 2499 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
To determine how Canadian physicians assess stroke risk in adults with atrial fibrillation and make therapeutic decisions around anticoagulation | 1 year

SECONDARY OUTCOMES:
To assess the adequacy of anticoagulation in treated patients | 1 year
To understand how new oral anticoagulants are incorporated into clinical practice | 1 year
To assess quality of life in patients with AF | 1 year
To evaluate how physicians select between rate and rhythm control options for AF | 1 year
To evaluate regional differences in care | 1 year
To compare management strategies between primary care physicians and cardiovascular specialists | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Milan K Gupta, MD, Principal Investigator — Canadian Collaborative Research Network; Andrew Ha, MD, Principal Investigator — Canadian Collaborative Research Network
Locations (1):
- CCRN, Brampton, Ontario, Canada

REFERENCES:
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Wann LS, Curtis AB, Ellenbogen KA, Estes NA 3rd, Ezekowitz MD, Jackman WM, January CT, Lowe JE, Page RL, Slotwiner DJ, Stevenson WG, Tracy CM, Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Kay GN, Le Heuzey JY, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann LS, Jacobs AK, Anderson JL, Albert N, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force. 2011 ACCF/AHA/HRS focused update on the management of patients with atrial fibrillation (update on Dabigatran): a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2011 Mar 15;123(10):1144-50. doi: 10.1161/CIR.0b013e31820f14c0. Epub 2011 Feb 14. No abstract available. PMID 21321155
- [Background] Dorian P, Guerra PG, Kerr CR, O'Donnell SS, Crystal E, Gillis AM, Mitchell LB, Roy D, Skanes AC, Rose MS, Wyse DG. Validation of a new simple scale to measure symptoms in atrial fibrillation: the Canadian Cardiovascular Society Severity in Atrial Fibrillation scale. Circ Arrhythm Electrophysiol. 2009 Jun;2(3):218-24. doi: 10.1161/CIRCEP.108.812347. Epub 2009 Mar 31. PMID 19808471
- [Background] Cairns JA, Connolly S, McMurtry S, Stephenson M, Talajic M; CCS Atrial Fibrillation Guidelines Committee. Canadian Cardiovascular Society atrial fibrillation guidelines 2010: prevention of stroke and systemic thromboembolism in atrial fibrillation and flutter. Can J Cardiol. 2011 Jan-Feb;27(1):74-90. doi: 10.1016/j.cjca.2010.11.007. PMID 21329865